CLINICAL TRIAL: NCT00390741
Title: Bone/Muscle Changes Following Hip Fracture in Older White Women
Brief Title: BHS4 - Bone/Muscle Changes Following Hip Fracture in Older White Women
Acronym: Hip4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jay S. Magaziner, Chair, Department Of Epidemiology & Public Health; Director, Center For Research On Aging, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-20834; NIA R37 AG09901
Record Dates: First submitted 2006-10-18; First posted 2006-10-20 (Estimated); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Hip Fracture
Keywords: hip fracture; bone mineral density; exercise
MeSH Terms: conditions — Hip Fractures; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Home-based exercise program
  Interventions: Behavioral: Exercise Plus Program
- 2 (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Exercise Plus Program — Those assigned to the treatment group were visited by an exercise trainer three times a week for the first two months of the study, two times per week during months three and four, one time per week during months five and six, two times a month during months seven and eight, and one time a month during months nine through twelve. During months seven through twelve of the study the trainer contacted the participant by telephone once each week during the weeks that he or she did not go the participants' home.
  Other Names: Exercise
  Arms: 1

SUMMARY:
The major goals of this study are:

1. To conduct an intervention development study to evaluate the feasibility of implementing an exercise intervention for reduction losses in bone mineral density, muscle mass, and strength, and clinically relevant aspects of functioning following a hip fracture, and to obtain preliminary tests of the effective ness of these interventions.
2. To evaluate the effect of home-based exercise intervention on bone metabolism.
3. To evaluate the effects of hip fracture on bone metabolism.
4. To evaluate the effects of exercise and hip fracture on hormonal regulators.
5. To evaluate the association between markers of bone metabolism hormone regulators, and BMD.
6. To separate out the effects of hip fracture on bone turnover from those of aging in persons with low bone mineral density.

DETAILED DESCRIPTION:
Hip fracture is a major public health problem, with striking consequences for the older patient, her family and the health care system. More than 350,000 persons over age 65 will fracture a hip in the United States during the coming year at an estimated annual cost of over $12 billion; by 2040, over 650,000 hip fractures will occur annually in this group. Between 18-33% of older hip fracture patients die within one year of their fracture, depending upon the specific population studied. Most surviving hip fracture patients experience reduced mobility and lose their ability to function independently. As many as 45% of those who are community dwelling at the time of their fracture are discharged to institutions post-hospitalization, and 15-25% remain institutionalized for a year post-fracture. Further, significant strain is observed in over a third of family caregivers as long as a year post-fracture. Depending upon the population studied and function being assessed, an estimated 25-75% of those who are independent before their fracture can neither walk independently nor achieve their previous level of independent living within a year following their fracture and 10- 20% of those who sustained a hip fracture can expect to have another osteoporotic fracture within two years.

This protocol consists of two components related to the recovery after hip fracture (described below):

EXERCISE INTERVENTION TRIAL. With few exceptions, which are restricted primarily to studies of comprehensive in-patient rehabilitation, little systematic attention has been given to evaluating strategies for improving functioning, bone, and muscle post-hip fracture. Strategies that have been shown to improve bone, muscle, and function in older persons who have not fractured a hip may be useful if applied to persons following hip fracture. Exercise is one of the strategies that have received considerable attention. Exercise training in older adults also has beneficial effects on bone density, muscle strength, and physical functioning, as well as cardiovascular fitness, and risk reduction for falls and fractures. An exercise program that combines weight-bearing and resistance exercises can increase bone mineral content in postmenopausal women. Little information is available on whether a home-based exercise program can be used to achieve similar benefits compared to a more structured, on-site exercise program. This issue is particularly relevant in older, frail women who have sustained a hip fracture because many are unable and unwilling to travel to exercise facilities.

Results of the studies of exercise are instructive of potential benefits for older persons following hip fracture. Most of the work to date has been restricted to relatively healthy, select samples of older persons who have been recruited into rigorously controlled randomized experiments. Hence, while they are efficacious in benefiting a select group of older persons, it is not known whether these interventions will be accepted by a frail older population which has become suddenly disabled by a hip fracture, nor is it known whether these interventions will be beneficial to this group which is losing bone, muscle and function at an accelerated rate.

Because losses in BMD following hip fracture place these women at greater rise of subsequent fracture and may delay or prevent full recovery of ambulatory ability, it is important to optimize fracture healing and prevent loss of bone. One therapeutic option for these patients that may be effective is to increase physical activity through exercise.

Despite these profound losses in function, bone, and muscle, we remain uncertain about the extent to which these losses can be attributed to the fracture, and only limited attention has been given to preventing such losses. In addition, we seek to understand the role of exercise in relation to bone metabolism and levels of hormones thought to regulate bone metabolism following a hip fracture. Elucidating these mechanisms will be valuable for understanding the effects of exercise on bone health. The purpose of this study is to take an intervention known to be beneficial in select populations, into the real world setting and apply to frail older persons who have become suddenly disabled by a hip fracture. It is essential to test the effectiveness of the intervention following a hip fracture.

With a waiver for authorization obtained at each hospital, the study nurse will do a chart review of hip fracture patients to determine study eligibility and then explain the study to the potential participant, obtain consent, and get baseline study measures within fifteen days of fracture. The project coordinator will notify the exercise trainers of which participants have been randomized to the treatment group, and the trainer will set up the first home visit.

After completing the baseline interview the participant will be assigned to one of two study groups. One group is the treatment group and one involves no treatment and are followed as usual care. Those assigned to the treatment group will be visited by an exercise trainer who will visit the participant three times a week for the first two months of the study, two times per week during months three and four, one time per week during months five and six, two times a month during months seven and eight, and one time a month during months nine through twelve. During months seven through twelve of the study the trainer will contact the participant by telephone once each week during the weeks that he or she does not go the participants' home.

Follow-up interviews, performance assessment, DEXA scans, ultrasound measurements (only for 34 participants) and blood draws will be done at two, six and twelve months following hip fracture. The baseline and follow-up interviews will last approximately two hours.

NON-HIP FRACTURE COMPARISON. Bone loss that occurs in older women is believed to result from uncoupling of bone remodeling. Despite the loss of BMD with aging, the cellular mechanisms for fracture healing appear to remain intact. Fracture healing can be divided into three phases: inflammatory, reparative, and remodeling. The first two phases are dependent primarily on the local trauma effects of the fracture and are completed within approximately five weeks; hence, exercise intervention would be expected to have little or no effect on these processes. The remainder of the approximately six-month duration of femoral neck fracture healing involves modeling and remodeling of the callus. Because skeletal loading may modulate remodeling, exercise should have an effect during this period. Even after completion of healing, mechanical factors are expected to continue to affect remodeling of the femur. Bone resorption, mediated by osteoclastic activity, is the first phase of a remodeling cycle. In the post-fracture context, in which both fracture debris removal and callus remodeling are ongoing, high levels of markers of resorption would be anticipated.

We will attempt to separate out the effects of hip fracture on bone turnover from those of aging in persons with low bone mineral density. Bone turnover of hip fracture patients receiving usual care will be compared to bone turnover in a similar group of women who have not fractured their hips (i.e., matched on age, ability to ambulate independently, and with low BMD).

ELIGIBILITY:
Inclusion Criteria:

* Hip fracture

Exclusion Criteria:

* Male
* Under 65 years old
* Non-surgical repair of hip fracture
* Non-community dwelling
* Fractured more than 72 hours before admission to the hospital
* Pathologic fracture
* Resides more than 70 miles from the hospital of admission
* Recent diagnosis (in past 6 months) of angina or myocardial infarction
* Myocardial infarction or stroke concurrent with hip fracture
* Diagnosis of ventricular arrhythmia, third degree heart block, atrial fibrillation or if vital signs equal heart less than 60 or greater than 100
* Active or suspected myocarditis or pericarditis in the past year
* Recent (within past 6 months) deep venous thrombosis or intracardiac thrombi
* Persistent pulmonary edema during hospitalization
* Poorly controlled blood pressure w/ resting systolic greater than 180 mm Hg or resting diastolic greater than 100 mm Hg (3 or more readings with 24- hour period)
* Presence of ventricular aneurysm
* Paget's Disease
* Diabetes--blood sugar consistently greater than 300
* Diagnosis of thyrotoxicosis or myxedema within past year
* Any diagnosis of hyperparathyroidism, hypoparathyroidism, or osteomalacia
* Parkinson's, multiple sclerosis, or ALS (Lou Gehrig's disease)
* New (past 6 months) onset seizure disorder or seizure within the past 6 months
* Diagnosis of schizophrenia
* Recent (within past 6 months) GI hemorrhage or bleeding
* Preadmission coumadin therapy
* Cirrhosis or end stage renal disease (ESRD)
* Advanced hepatitis, AIDS, or endocarditis
* Cancer with metastases, or cancer under active treatment (chemotherapy with cytotoxic agents) other than non-melanomic skin cancers
* Current diagnosis of chronic alcohol abuse
* Preadmission narcotic use or preadmission benzodiazepine use more than 1 dose or tablet a day
* Required human assistance to walk prior to fracture
* Prior fracture
* Chest pains when climbing a flight of stairs, while walking on level ground, or at rest prior to the hip fracture
* Use of supplemental oxygen prior to fracture
* Other (Non-English speaking, severe blindness, paraplegia, hemiplegia
* Mini-Mental Status Exam score less than 20

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 170 (Actual)
Dates: Start 1998-10; Primary Completion 2004-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Self-efficacy | 2, 6, and 12 months post hip fracture
Exercise behavior and activity | 2, 6, and 12 months post hip fracture
Subjective reporting of exercise | 2, 6, and 12 months post hip fracture

SECONDARY OUTCOMES:
Compliance | 2, 6, and 12 months post hip fracture
Change in BMD | 2, 6, and 12 months post hip fracture
Lower extremity function | 2, 6, and 12 months post hip fracture
Falls | 2, 6, and 12 months post hip fracture
Time to weight bearing | 2, 6, and 12 months post hip fracture
Dietary intake | 2, 6, and 12 months post hip fracture

CONTACTS AND LOCATIONS:
Overall Officials: Jay Magaziner, Ph.D., MSHyg, Principal Investigator — University of Maryland, Baltimore
Locations (3):
- United States (3):
  - Union Memorial Hospital, Baltimore, Maryland
  - Northwest Hospital Center, Randallstown, Maryland
  - St. Joseph's Hospital, Towson, Maryland

REFERENCES:
- [Derived] Orwig DL, Hochberg M, Yu-Yahiro J, Resnick B, Hawkes WG, Shardell M, Hebel JR, Colvin P, Miller RR, Golden J, Zimmerman S, Magaziner J. Delivery and outcomes of a yearlong home exercise program after hip fracture: a randomized controlled trial. Arch Intern Med. 2011 Feb 28;171(4):323-31. doi: 10.1001/archinternmed.2011.15. PMID 21357809